CLINICAL TRIAL: NCT02979509
Title: Multi-center Prospective Evaluation of the Diagnostic Yield of Endoscopic Ultrasound-Guided Tissue Sampling
Brief Title: Evaluation of Diagnostic Yield of EUS-Guided Tissue Sampling
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Borland Groover Clinic, Jacksonville, FL (Unknown); Northwestern University, Chicago, IL (Unknown); Mayo Clinic (Other); Montefiore Medical Center, Bronx, NY (Unknown); Columbia University (Other); Johns Hopkins University (Other); New York University, New York, NY (Unknown); Yale University (Other); Geisinger Medical Center, Danville, PA (Unknown); Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600783
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Gastroenterology; Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic ultrasound- (EUS) guided tissue sampling: All patients scheduled to undergo EUS with tissue sampling (TS) as medically indicated will be considered for the study. Patients in whom EUS-TS is considered as part of their standard medical care will be offered to participate in this study.
  Interventions: Other: Endoscopic ultrasound- (EUS) guided tissue sampling

INTERVENTIONS:
Other: Endoscopic ultrasound- (EUS) guided tissue sampling — EUS- guided tissue sampling of solid and/or cystic pancreatic and non-pancreatic lesions as part of their medical care.
  Other Names: EUS-TS

SUMMARY:
All patients will receive standard medical care and no experimental interventions will be performed. Endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) is a well-established procedure commonly used for the investigation of lesions within or adjacent to the gastrointestinal (GI) lumen (i.e. pancreas, liver, mediastinal masses, left adrenal gland, lymph nodes, and subepithelial lesions). EUS-guided tissue sampling has been commonly performed with different size and types of aspiration and core biopsy needles.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) is a well-established procedure commonly used for the investigation of lesions within or adjacent to the gastrointestinal (GI) lumen (i.e. pancreas, liver, mediastinal masses, left adrenal gland, lymph nodes, and subepithelial lesions). EUS-guided tissue sampling has been commonly performed with different size and types of aspiration and core biopsy needles. More recently, a novel through-the-needle microforceps has been introduced. The MorayTM microforceps fits through a 19-gauge FNA needle and allows targeted tissue sampling under EUS visualization.

Aim - To prospectively evaluate the safety and diagnostic yield of the through-the-needle microforceps for pancreatic and non-pancreatic solid, cystic and mixed solid/cystic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Patients referred for EUS-guided tissue sampling for lesions (i.e. pancreas, liver, mediastinal masses, left adrenal gland, lymph nodes, and subepithelial lesions).
3. Target lesion should be ≥ 15 mm in size (long axis).

Exclusion Criteria:

1. Any contraindication to performing endoscopy
2. Unable to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include all patients who are scheduled to undergo EUS-guided tissue sampling as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Overall diagnostic yield of EUS-TS | 2 months

SECONDARY OUTCOMES:
Diagnostic Yield of EUS-guided tissue sampling solid lesions | 2 months
Diagnostic Yield of EUS-guided tissue sampling cystic lesions | 2 months
Diagnostic yield of EUS-TS using through-the-needle micro forceps | 2 months
Diagnostic yield of EUS-TS using fine-needle aspiration | 2 months
Diagnostic yield of EUS-TS using core biopsy needle | 2 months
Rate of adverse events associated with EUS-TS | 48 hours
  Adverse events defined based on previously established criteria by the American Society of Gastrointestinal Endoscopy (ASGE)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Computer-based files will only be made available to personnel involved in the study through the use of access privileges, passwords and encryption. The prospectively maintained database will be constructed with the Research Electronic Data Capture software.

REFERENCES:
- [Derived] Yang D, Trindade AJ, Yachimski P, Benias P, Nieto J, Manvar A, Ho S, Esnakula A, Gamboa A, Sethi A, Gupte A, Khara HS, Diehl DL, El Chafic A, Shah J, Forsmark CE, Draganov PV. Histologic Analysis of Endoscopic Ultrasound-Guided Through the Needle Microforceps Biopsies Accurately Identifies Mucinous Pancreas Cysts. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1587-1596. doi: 10.1016/j.cgh.2018.11.027. Epub 2018 Nov 22. PMID 30471456